CLINICAL TRIAL: NCT02189083
Title: A Double-blind, Randomized, Two-dose Trial of Tumor-shrinking Decoction (TSD), a Chinese Medicine Preparation in Patients With Symptomatic Uterine Fibroids
Brief Title: Study of Tumor-shrinking Decoction (TSD) to Treat Symptomatic Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU-SCM-TSD2014; HMRF-11121841 (Other Grant/Funding Number: Health and Medical Research Fund (HMRF))
Record Dates: First submitted 2014-05-14; First posted 2014-07-14 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2014-07

CONDITIONS: Leiomyoma
Keywords: Leiomyoma; Medicine, Chinese Traditional; Randomized Controlled Trial
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose TSD (Experimental): Subjects in this arm receive high dose (217 g/day) TSD for 16 weeks.
  Interventions: Drug: TSD
- Low dose TSD (Active Comparator): Subjects in this arm receive low dose (69 g/day) TSD for 16 weeks.
  Interventions: Drug: TSD

INTERVENTIONS:
Drug: TSD — TSD is composed of 15 individual Chinese medicines: Astragalus Membranaceus, Semen Coicis, Poria, Curcuma longa L, and Fritillaria Thunbergii Miq, Cassia twig, Pollen typhae, Resina draconis, Lithospermum erythrorhizon, Halloysitum Rubrum, Rhizoma Corydalis processed with vinegar, Hirudo, Calcined corrugated sub , Oyster Shell and Laminaria Japonica Aresch.
  High dose (127g) or Low dose (69g) TSD decoction boiled as 200ml per bag; 2 bags per day, 6 days per week; Orally in-take one bag of TSD decoction in morning and another in evening after meal; The whole treatment lasts for 16 weeks.
  Other Names: Tumor-shrinking Decoction, Chinese medicine preparation

SUMMARY:
On the basis of empirical evidence and clinical practice, the investigators have developed a formula called Tumor-shrinking Decoction (TSD) used in the treatment of uterine fibroids (UFs). The investigators preliminary clinical observation has demonstrated the benefits of TSD in improving UFs.

TSD is composed of 15 individual Chinese medicines: Astragalus Membranaceus, Semen Coicis, Poria, Curcuma longa L, and Fritillaria Thunbergii Miq, Cassia twig, Pollen typhae, Resina draconis, Lithospermum erythrorhizon, Halloysitum Rubrum, Rhizoma Corydalis processed with vinegar, Hirudo, Calcined corrugated sub , Oyster Shell and Laminaria Japonica Aresch.

It is hypothesized that TSD can effectively reduce the fibroid size and improve the symptoms associated with UFs and the greater anti-tumor potency of TSD is associated with higher therapeutic doses.

To test this hypothesis, one 16-week, double-blind, randomized, two-dose trial will be conducted in patients with symptomatic UFs to determine whether the high dose (217 g/day) of TSD could produce significantly greater effects in reducing the fibroid size and improving its related symptoms and biochemical profiles compared to the lower dose (69 g/day).

DETAILED DESCRIPTION:
Numerous Chinese medicine preparations have been shown to possess therapeutic potential in relieving uterine fibroids (UFs) symptoms and shrinking the volume of fibroids without significant adverse effects, although the clinical efficacy needs to be further confirmed with rigorously designed.On the basis of empirical evidence and clinical practice, the investigators have developed a formula called Tumor-shrinking Decoction (TSD) used in the treatment of UFs. The investigators preliminary clinical observation has demonstrated the benefits of TSD in improving UFs.

TSD is composed of 15 individual Chinese medicines. According to traditional Chinese medicine (TCM) doctrine, most UFs are developed due to the deficiency of vital energy and the stasis of blood, resulting in the formation of pathological massive tissues. Individual Chinese medicines constituting TSD can be classified into three classes based on TCM-defined pharmacological actions: (i) Tonifying qi and resolve phlegm: Astragalus Membranaceus, Semen Coicis, Poria, Curcuma longa L, and Fritillaria Thunbergii Miq; (ii) Resolve stasis, stopping bleeding and relieve pain: Cassia twig, Pollen typhae, Resina draconis, Lithospermum erythrorhizon, Halloysitum Rubrum, Rhizoma Corydalis processed with vinegar; and (iii) Softening hardness and dissipate binds: Hirudo, Calcined corrugated sub , Oyster Shell and Laminaria Japonica Aresch.

Indeed, the investigators previous studies of cultured cells and animals have revealed that TSD robustly inhibits fibroid cell growth and proliferation. The investigators therefore hypothesize that TSD can effectively reduce the fibroid size and improve the symptoms associated with UFs and the greater anti-tumor potency of TSD is associated with higher therapeutic doses.

To test this hypothesis, one 16-week, double-blind, randomized, two-dose trial will be conducted in patients with symptomatic UFs to determine whether the high dose (217 g/day) of TSD could produce significantly greater effects in reducing the fibroid size and improving its related symptoms and biochemical profiles compared to the lower dose (69 g/day).

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women aged 18 to 52 years; and
2. have a primary diagnosis of symptomatic UFs based on clinical symptoms; and
3. MRI examination as defined in the International Classification of Diseases (10th edition).

Exclusion Criteria:

1. Unstable medical conditions such as serious cardiovascular diseases;
2. With severe neuropsychiatric disorders;
3. Combined with adenomyosis or other tumors;
4. On treatment with Chinese medicine or other natural products in the previous 3 months;
5. With an allergic history of herbal medicine; or
6. Being pregnant and lactating women and those who currently use contraception.

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in the symptom severity score of Uterine Fibroid Symptom and Quality of Life questionnaire (UFS-QOL) from Baseline to 6 months | Baseline and once per month thereafter; Up to 6 months
  UFS-QOL consists of 37 items to assess the severity of UFs-related symptoms and the quality of life of patients.

SECONDARY OUTCOMES:
Change of clinical response from baseline on the the health-related quality of life of transformed UFS-QOL score | Baseline and once per month thereafter; Up to 6 months
  The secondary clinical outcome is the clinical response that is defined as a ≥30% baseline-to-endpoint reduction on the symptom severity of transformed UFS-QOL score.
Imaging outcomes | Baseline, 5th month
  Imaging outcomes will be examined at baseline and endpoint using magnetic resonance imaging (MRI) scan to determine the number, size and density of the uterine fibroids.
Serum concentrations of estrogen and follicle-stimulating hormone | Baseline, 5th month
  two blood samples will be collected from each patient at baseline and at the end of the study, respectively. The collection of blood will be conducted between 08:00 and 09:00 before meal. Sera will be separated and stored at -20ºC until assayed. Serum concentrations of estrogen, progesterone and follicle-stimulating hormone will be measured using chemiluminescent immunoassay (CLIA).

OTHER OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 6 months
  Adverse events will be closely monitored at each visit. All adverse events, reported, elicited or observed, will be recorded on case report form, including the date and time of onset, duration, severity, relationship to study drug, and action taken.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Meng, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Chinese Medicine, University of Hong Kong, Hong Kong, China

REFERENCES:
- [Result] Lu J, Meng W. Clinical observation 45 cases of Yiqi Huayu treatment for uterine fibroids. Gansu TCM. 2008a;6:44-46
- [Result] Lu J, Meng W. Clinical Observation of " Hualiu Recipe" in Treating 302 Cases of Hysteromyoma with Qi- Deficiency and Blood- Stasis Syndrome. Shanghai Traditional Chinese Medicine. 2008b;3:49-51
- [Result] Meng W, Ma B. Three drugs on cultured uterine leiomyoma cell proliferation and apoptosis, and regulatory factors. Traditional Chinese. 2003;21:2046-2048
- [Result] Meng W. Zhao W. Effects of methods of invigorating qi and dissolving stasis on the expression of proliferating and apoptosis of cultured human uterine leiomyoma cells. Chinese archives of traditional Chinese medicine. 2008(2);238-240
- [Result] Tan L, Meng W, Zhang TT. [Predisposing factors of hysteromyoma and effect of hualiu recipe on it]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2011 May;31(5):635-8. Chinese. PMID 21812264
- See also: American Society of Reproductive Medicine Patient Booklet: Uterine Fibroids — http://www.asrm.org/FactSheetsandBooklets/